CLINICAL TRIAL: NCT01799668
Title: Therapists' Preferences for Client Characteristics and Their Influence on the Therapeutic Alliance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Ahud Sternberg, MD, Hillel Yaffe Medical Center
Other Study IDs: 0001-13 HYMC
Record Dates: First submitted 2013-02-10; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Diagnosis, Psychiatric; Outpatient Followup of Psychiatric Problem
Keywords: Psychotherapy; Preferences
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
The research will examine psychotherapists' preferences for theoretical client characteristics, such as age, gender, personality characteristics and symptoms. The research will also examine the preferences' influence on the therapeutic alliance, from the therapist's and the client's point of view.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients over the age of 18,
* Hebrew speakers,
* Not in a psychotic state.

Exclusion Criteria:

* Psychotic state,
* Under the age of 18,
* Not qualified to answer the questions,
* Don't speak any Hebrew at all.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients in the psychiatric department
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Positive correlation between preferences- characteristics match and therapeutic alliance. | 5 weeks
  The match between therapists' preferences ant their client's characteristics will correlate positively with the measures of therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Ella Landa, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel